CLINICAL TRIAL: NCT03695406
Title: Mind Body Program for Fear of Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017P000168
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Cancer Survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind-Body Group Intervention (Experimental)
  Interventions: Behavioral: Mind-Body Program for Fear of Recurrence

INTERVENTIONS:
Behavioral: Mind-Body Program for Fear of Recurrence — An adapted protocol of the Relaxation Response Resiliency Program, a manualized, group-based, multimodal mind body program. Protocol adaptation includes refinement of content and study procedures to target fear of cancer recurrence (FCR) among adult cancer survivors.

SUMMARY:
This is a pilot feasibility study of a group-based, mind body intervention for managing stress and fear of recurrence and promoting resiliency among adult cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a history of breast, lung, colorectal, hematologic, prostate, melanoma, or gynecological cancer (by medical record and/or self-report)
2. Completion of primary cancer treatment (radiation, surgery, and/or chemotherapy) between 3 to 30 months ago
3. Ages 18 and older (by medical record and/or self-report)

Exclusion Criteria:

1. Self-reported inability to speak and write in English
2. Concurrent participation in weekly, group-based psychosocial or mind-body programs
3. Serious mental illness (by medical record and/or self-report) as defined by history of suicidality, psychosis, and/or psychiatric hospitalization in the past year.
4. Inability to travel to necessary study visits
5. No e-mail address to access online assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Feasibility (i.e., retention at initial follow-up assessment) | Through study completion (approximately 5 months)
  The primary metric for assessing Feasibility will be retention at the initial follow-up assessment. Reasons for ineligibility, refusal, or dropping out will be measured.
Acceptability | During intervention group sessions (approximately 2 months)
  The primary metric for assessing Acceptability will be a five-item, investigator developed self-report questionnaire. Following each study session, participants will be asked to rate (1=not at all to 5=very much) the enjoyableness, convenience, helpfulness, relevancy, odds of future use, and overall satisfaction of the session.

SECONDARY OUTCOMES:
Fear of Cancer Recurrence | Baseline, 8 weeks (Post-intervention), 1 month follow-up, 3 months follow-up
  Fear of Cancer Recurrence Inventory. Validated self-report measure of fear of cancer recurrence. 42 items across 7 subscales (triggers, severity, psychological distress, coping strategies, functioning impairments, insight, and reassurance). Higher scores indicate more fear of recurrence. Severity subscale score ≥16 indicates elevated FCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medial Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall DL, Park ER, Cheung T, Davis RB, Yeh GY. A Pilot Mind-Body Resiliency Intervention Targeting Fear of Recurrence among Cancer Survivors. J Psychosom Res. 2020 Oct;137:110215. doi: 10.1016/j.jpsychores.2020.110215. Epub 2020 Aug 10. PMID 32818720